CLINICAL TRIAL: NCT01529021
Title: Reducing Children's Distress Towards Flu Vaccinations
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tanya Beran, Associate Professor, University of Calgary
Other Study IDs: E 23795
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Children's Distress During Flu Vaccination
Keywords: Pain management; vaccination; immunization; pediatric; robotics; human-robot interaction
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- humanoid robot distration: The robot NAO, academic edition (Aldebaran Robotics) was used in this study. Some of its features include an on-board fully programmable computer CPU: x86 AMD Geode with 500 MHz, 256 MB SDRAM and 1 GB flash memory, WiFi (802.11g) and Ethernet, two cameras with up to 30 frames per second, two hands with self adaptive gripping abilities, force sensitive sensors on its arms and feet to perceive contact with objects, Light Emission Diodes in its eyes and body, four microphones to identify the source of sounds, and two loud speakers for communication where tone and voice pitch can be modified in real-time. It runs on a native Linux Operating system platform and can be programmed using a proprietary SDK called NaoQi, or in C, C++, Ruby and Urbi, which makes it compatible with other robot simulators such as Microsoft Robotics Developer Studio.
- control: standard care procedures were used during the vaccination

SUMMARY:
Millions of children in North America receive an annual flu vaccination, many of whom are at risk of experiencing severe distress. Children frequently use technologically advanced devices such as computers and cell phones. Based on this familiarity, the investigators introduced another sophisticated device - a humanoid robot to- interact with children during their vaccination. The investigators hypothesized that these children would experience less distress than children who did not have this interaction.

DETAILED DESCRIPTION:
57 children (30 male; age, mean + SD: 6.87 + 1.34 years) were randomly assigned to a vaccination session with a nurse who used standard administration procedures, or with a robot who was programmed to use cognitive-behavioral strategies with them while a nurse administered the vaccination. Measures of distress were completed by children, parents, nurses, and researchers.

ELIGIBILITY:
Inclusion Criteria:

* ages 5-9 years,
* boys and girls

Exclusion Criteria:

* children with pervasive developmental disability

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children in the general public and from hospital ages 5-9 years
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale-Revised | 5 mins before and immediate after vaccination
  The Faces Pain Scale-Revised was administered to children and their parents while in the waiting room and after consent was signed. Once this questionnaire and consent were completed, the parent and child entered the vaccination room for the vaccination. As soon as the vaccination was completed, the Faces Pain Scale-Revised was re-administered.

SECONDARY OUTCOMES:
Behavioral Approach-Avoidance Distress Scale | one week after vaccination was administered
  The Behavioral Approach-Avoidance Distress Scale was used by researchers one week after the data collection phase was completed while reviewing the videos.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Beran, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Beran TN, Ramirez-Serrano A, Vanderkooi OG, Kuhn S. Reducing children's pain and distress towards flu vaccinations: a novel and effective application of humanoid robotics. Vaccine. 2013 Jun 7;31(25):2772-7. doi: 10.1016/j.vaccine.2013.03.056. Epub 2013 Apr 24. PMID 23623861